CLINICAL TRIAL: NCT06634615
Title: The Effect of Patient Education and in the Operating Room Family Interview Practices on Patient Outcomes Using Virtual Reality in Cholecystectomy Patients: A Randomized Controlled Trial
Brief Title: The Effect of Patient Education and in the Operating Room Family Interview Practices on Patient Outcomes Using Virtual Reality in Cholecystectomy Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Çağla Islattı Mutlu, Research Assistant, Nurse, Marmara University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 09.2024.646
Record Dates: First submitted 2024-10-08; First posted 2024-10-10 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2024-09

CONDITIONS: Cholecystectomy, Laparoscopic; Virtual Reality; Patient Education; Family Interviews; Operating Room; Anxiety; Stress; Sleep Quality; Patient Satisfaction; Patient Outcomes
Keywords: Cholecystectomy; Virtual Reality; Patient Education; Operating Room Family Interview; Patient Outcomes; Anxiety; Stress; Sleep Quality; Patient Satisfaction
MeSH Terms: conditions — Anxiety Disorders; Sleep Initiation and Maintenance Disorders; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: There are three groups in the study: a patient education group with virtual reality glasses, a patient education group with virtual reality glasses and video family interview, and a control group without education and/or interview.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Education (Experimental): Patients in the education group will be shown a patient education video about the laparoscopic cholecystectomy operation with virtual reality glasses on the day of hospitalization.
  Interventions: Other: VR patient education video
- Education+Interview (Experimental): Patients in the education+interview group will be shown a patient education video about the laparoscopic cholecystectomy operation with virtual reality glasses on the day of hospitalization. Patients in the education group will be shown a patient education video on laparoscopic cholecystectomy surgery with virtual reality glasses on the day of admission to the hospital. When patients are taken to the operative waiting area, virtual reality glasses will be put on and a 5-minute video family meeting will be initiated with the patient's relative(s).
- Control (No Intervention)

INTERVENTIONS:
Other: VR patient education video — The educational video is created by converting the information provided by the service nurses into a video when the patient is admitted to the ward for surgery. The video will show a 2-3 minute animation of a nurse giving information. In a patient room, the service nurse will come to the newly admitted patient and explain the concept of cholecystectomy, the reasons for removing the gallbladder, how laparoscopic cholecystectomy is performed, the advantages of laparoscopic surgery compared to open surgery, the preparation process before and on the day of surgery, the conditions to be monitored after surgery, the importance of nutrition and fluid intake, defecation, the importance of early mobilization and discharge.
  Arms: Education
Other: VR family interview — Patients will have a 5-minute video call with their families in a 360° designed home environment using virtual reality glasses in the operating room waiting area.

SUMMARY:
This study was planned to be a randomized controlled experimental study to determine the effect of patient education and family interview practices using virtual reality on stress intensity, anxiety and information need levels, sleep quality and satisfaction with the preparation process for surgery in cholecystectomy patients. The main questions it aims to answer are:

* Is there a significant difference in stress intensity, anxiety, and information need levels between patients who received and did not receive patient education with VR glasses in the ward before cholecystectomy surgery?
* Is there a significant difference in stress intensity and anxiety levels between patients who received and did not receive video family interviews with VR glasses in the operative waiting area before cholecystectomy surgery?
* Is there a significant difference in stress intensity, anxiety, and sleep quality levels at discharge of groups that received different VR interventions?
* What is the postoperative sleep quality of patients with low preoperative anxiety levels?
* What is the satisfaction of patients who received VR with the surgery preparation process? The patients participating in the study will be numbered according to the order of hospitalization and assigned to one of the control, education, education+interview groups in accordance with the randomization list. Face-to-face communication will be established with each patient in the ward on the day of hospitalization, in the preoperative waiting area when they come to the operating room and in the ward on the day of discharge. Depending on the groups in which the patients are included, they will be shown an educational video using virtual reality goggles and/or will be allowed to meet with their families. No application will be made to the control group and the ward routine will continue.

DETAILED DESCRIPTION:
Virtual reality (VR) is an interactive field that offers sensory experiences such as three-dimensional vision, touch and hearing, allowing people to dive into the virtual world and feel that they are in a different environment. In healthcare services, it is seen that the effect of virtual reality technology on various patient outcomes has been examined by watching nature videos, training, exercise applications, museum tours with music and games. This study was planned to be a randomized controlled experimental study to determine the effect of patient education and family interview practices using virtual reality on stress intensity, anxiety and information need levels, sleep quality and satisfaction with the preparation process for surgery in cholecystectomy patients. G*Power (v3.1.9.7) program was used to determine the sample size in the study and considering possible losses, it was decided to include a total of 60 patients, 20 in each group.

During the data collection process, it is planned to include a total of six patients in the preliminary pilot application, two from the education group, two from the education+interview group, and two from the control group, for the comprehensibility and usability of the forms. Patients who have undergone preliminary application will not be included in the study. The patients participating in the study will be numbered according to the order of hospitalization and assigned to one of the control, education, education+interview groups in accordance with the randomization list. Face-to-face communication will be established with each patient in the ward on the day of hospitalization, in the preoperative waiting area when they come to the operating room and in the ward on the day of discharge. The first interview with the patients will be held in the patient room in the ward. During this interview, the patients will be invited to the study and the research will be explained. Informed voluntary consent will be obtained from the patients who agree to participate in the study. Depending on the groups in which the patients are included, they will be shown an educational video using virtual reality goggles and/or will be allowed to meet with their families. Data will be collected with the Introductory Information Form, Visual Analog Scale for Stress, Amsterdam Preoperative Anxiety and Information Scale (APAIS), Richards Campbell Sleep Scale (RCBS), Virtual Reality Evaluation Form and Visual Analog Scale for Satisfaction. Oculus Quest 2 VR glasses will be used as a virtual reality application tool in the study.

The virtual family meeting will be initiated through the meeting link shared with the patients relative, and VR glasses and computer connection will be provided with the BigScreen computer application. Patients have a video call with their family in a 360° designed home environment. The conversations are easily transmitted thanks to the internal speaker and microphone in the VR glasses. In order to adjust the patients viewing angle, to provide guidance when needed, and to monitor communication, the image the patient sees in the VR glasses will be monitored with the Meta Quest program installed on the researchers mobile phone. The training video is a 2-3 minute animated video with visual and auditory elements and includes the ward nurse coming to the newly admitted patient in a patient room and giving information. In order to prevent infection, after each patients use, the supporting pads, straps, and lenses of the virtual reality glasses will be disinfected with cleaner and allowed to dry. It will be kept in its own box and offered to the other patients use.

In the first phase of the study with the patients in the control group, the data collection tools including the Introductory Information Form, the Visual Analog Scale for Stress, the Amsterdam Preoperative Anxiety and Information Scale (APAIS) and the Richard-Campbell Sleep Scale (RCS) will be filled in on the day of admission. No intervention will be applied to the patients and routine procedures will continue. After 30 minutes, the patient will be asked to fill in the Visual Analog Scale for Stress and the Amsterdam Preoperative Anxiety and Information Scale (APAIS) again. In the second phase of the study, when the patients are taken to the preoperative waiting area of the operating room, the data collection tools including the Visual Analog Scale for Stress and the Amsterdam Preoperative Anxiety and Information Scale (APAIS) will be filled in. At the end of the period in which the patient waits to be taken to the operation, the patient will be asked to fill in the Visual Analog Scale for Stress and the Amsterdam Preoperative Anxiety and Information Scale (APAIS) again. In the final phase of the study, the Stress visual analog scale, Amsterdam preoperative anxiety and information scale (APAIS), Richard-Campbell sleep scale (RCUS) and Satisfaction visual analog scale will be filled in the patient room before discharge on the morning of the first postoperative day.

In the first phase of the study, the patients in the patient education group will first fill out the data collection tools including the Introductory Information Form, Stress visual analog scale, Amsterdam preoperative anxiety and information scale (APAIS) and Richard-Campbell sleep scale (RCUS) on the day of admission. Then, a patient education video about laparoscopic cholecystectomy operation will be watched with virtual reality glasses. 30 minutes after watching the education video, patients will be asked to fill out the Stress visual analog scale and Amsterdam preoperative anxiety and information scale (APAIS) again. In the second phase of the study, when the patients are taken to the preoperative waiting area of the operating room, the Stress visual analog scale and Amsterdam preoperative anxiety and information scale (APAIS) will be filled in the data collection tools including the Stress visual analog scale and Amsterdam preoperative anxiety and information scale (APAIS). At the end of the waiting period for the patient to be taken to the operation, they will be asked to fill out the Stress Visual Analog Scale and Amsterdam Preoperative Anxiety and Information Scale (APAIS) again. In the last stage of the study, on the morning of the first post-operative day, before discharge, the patient will be asked to fill out the data collection forms including the Stress Visual Analog Scale, Amsterdam Preoperative Anxiety and Information Scale (APAIS), Richard-Campbell Sleep Scale (RCUS), Virtual Reality Evaluation Form and Satisfaction Visual Analog Scale in the patient room.

In the first stage of the study, the patients in the Education + Interview group will first fill out the data collection tools including the Introductory Information Form, Stress Visual Analog Scale, Amsterdam Preoperative Anxiety and Information Scale (APAIS) and Richard-Campbell Sleep Scale (RCUS) on the day of admission. Then, a patient education video regarding laparoscopic cholecystectomy operation will be watched with virtual reality glasses. After watching the training video, patients will be asked to fill out the Stress Visual Analog Scale and Amsterdam Preoperative Anxiety and Information Scale (APAIS) again 30 minutes later. In the second phase of the study, when patients are taken to the preoperative waiting area, data collection tools including the Stress Visual Analog Scale and Amsterdam Preoperative Anxiety and Information Scale (APAIS) will be filled out. After the patient is put on virtual reality glasses and his/her vision is adjusted, a video family interview will be initiated. After the 5-minute virtual visit with the patients relative(s), the interview will be concluded and the Stress Visual Analog Scale, Amsterdam Preoperative Anxiety and Information Scale (APAIS) will be filled out again. In the last phase of the study, data collection forms including the Stress Visual Analog Scale, Amsterdam Preoperative Anxiety and Information Scale (APAIS), Richard-Campbell Sleep Scale (RCUS), Virtual Reality Evaluation Form and Satisfaction Visual Analog Scale will be filled out in the patients room before discharge on the morning of the first postoperative day.

ELIGIBILITY:
Inclusion Criteria:

* Patients who volunteered to participate in the study,
* who were 18 years of age or older,
* who would undergo elective laparoscopic cholecystectomy surgery,
* who had no vision, hearing and communication problems,
* whose relatives had a smartphone and internet connection,
* whose stress intensity was higher than 3 points (between 1-10 points) met the inclusion criteria.

Exclusion Criteria:

* Patients with complaints of dizziness,
* psychiatric disorders,
* persistent sleep problems were excluded from the study.
* Patients who voluntarily left the study,
* interrupted the family video call with VR,
* felt discomfort during VR application,
* developed any allergy to the goggle material,
* filled out the data collection forms incompletely and/or incorrectly will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-05 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Stress | On the day of hospitalization, during the first interview with the researcher and 30 minutes later; When arriving in the operating room waiting area and before going to the operation; On the morning of the first post-operative day, before discharge.
  It is an 11-step scale ranging from 0-I am not stressed at all, to 10-I am very stressed, on a 10 cm ruler to assess the stress intensity of patients. The ruler shows that the stress level increases as it goes from 0 to 10.
Anxiety and need for information | On the day of hospitalization, during the first interview with the researcher and 30 minutes later; When arriving in the operating room waiting area and before going to the operation; On the morning of the first post-operative day, before discharge.
  Total scale score is min. 6 and max. 30. High scores are associated with high anxiety levels and desire for information.
Sleep | On the day of hospitalization, during the first interview with the researcher and on the morning of the first postoperative day before discharge.
  Each item of the scale is evaluated and answered on a chart ranging from 0 to 100. A score between "0-25" from the scale indicates very poor sleep, and a score between "76-100" indicates very good sleep.
Satisfaction with the preparation process for surgery | Post-op 1st day morning before discharge.
  It is an 11-step scale ranging from 0-Not satisfied at all, 10-Very satisfied on a 10 cm ruler. The ruler shows that the level of satisfaction increases as it goes from 0 to 10.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University Pendik Training and Research Hospital Prof. Dr. Asaf Ataseven Additional Service Building, Istanbul, Turkey (Türkiye)